CLINICAL TRIAL: NCT02984397
Title: Proof of Concept Trial to Test the Efficacy of Treatment With Ketotifen on Pain Sensitivity and Association Between Level of Activity and Reactivity of White Blood Cells and Pain Sensitivity in Teenagers With Chronic Widespread Pain
Brief Title: Chronic Widespread Pain and White Blood Cell Activation
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Collaborators: The Louise And Alan Edwards Foundation (Unknown)
Responsible Party: Principal Investigator, Pablo Ingelmo, Associate Professor, Department of Anesthesia; Director, Chronic Pain Service (Pediatric), Montreal Children's Hospital, McGill University Health Centre/Research Institute of the McGill University Health Centre
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 15-207-MUHC
Record Dates: First submitted 2016-12-02; First posted 2016-12-06 (Estimated); Last update posted 2020-02-20 (Actual); Status verified 2020-02

CONDITIONS: Widespread Chronic Pain
Keywords: pain; ketotifen; pediatric; mast cell
MeSH Terms: conditions — Chronic Pain; Pain | interventions — Ketotifen; Standard of Care

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- KF group (Experimental): In each study visit, patients will receive enough pills for the next month. At the first visit, patients receiving ketotifen (KF) will receive four vials sequentially numbered (1 to 4) containing enough pills for one week each, and will be instructed by the clinician and by the pharmacist to use vial 1 for the first week (0.5 mg of KF BDI), vial 2 for the second week (1mg of KF BDI), vial 3 for the third week (2 mg of KF BDI), and vial 4 for the fourth week (3mg of KF BDI). As for weeks 4, 8 and 12 visits, patients treated with KF will receive four equal vials containing enough pills for one week each (3 mg of KF BDI)
  Interventions: Drug: Ketotifen Fumarate
- Placebo group (Placebo Comparator): Patients participating in the placebo group will also receive sequentially numbered vials at the first visit. Similarly, patients taking placebo will also receive four equal vials of pills on the next visits.
  Interventions: Drug: Placebo
- SOC (Active Comparator): Standard of care - patients who refuse to participate in the study but allow us to compare their clinical data to that of participants of the study
  Interventions: Other: Standard of Care

INTERVENTIONS:
Drug: Ketotifen Fumarate — Ketotifen is a second-generation noncompetitive H1-antihistamine and mast cell stabilizer. It is most commonly sold as a salt with fumaric acid, ketotifen fumarate, and is available in two forms. In its ophthalmic form, it is used to treat allergic conjunctivitis, or the itchy red eyes caused by allergies. In its oral form, it is used to prevent asthma attacks.
  Other Names: Zaditen
  Arms: KF group
Drug: Placebo
  Arms: Placebo group
Other: Standard of Care
  Arms: SOC

SUMMARY:
Our goal is to conduct a proof-of-concept trial to test the efficacy of KF treatment in adolescents with severe CWP not responding to the standard of care (SOC) treatment program in a multidisciplinary tertiary care chronic pain clinic. The changes associated to the interventions (KF or placebo) will be quantified using the Patients' Global Impression of Change (PGIC) scale after 16 weeks of treatment. Secondary, we aim to evaluate the effects of KF on the pain sensitivity, physical and emotional functioning, and we will also explore the potential biological underlying mechanisms.

DETAILED DESCRIPTION:
We have designed a proof-of-concept (POC) trial composed of three arms. The first two arms will be a randomized, controlled, double-blind, parallel-group study, designed to assess the potential efficacy of KF for the treatment of pain and associated symptoms in adolescent with CWP. The third arm will consists of assessing standard of care (SOC) data from patients who do not wish to participate in the study, but agree to allow us to use their SOC data to be compared with that of patients participating in the study. This arm will help to evaluate the potential beneficial effect of being part of the study ("placebo" effect) receiving a new treatment for a condition where the SOC have limited success rate.

ELIGIBILITY:
Inclusion Criteria:

* Female and male adolescents aged between 14 to 18 years old;
* For female adolescents of child bearing potential: negative serum pregnancy test at base line screening;
* For female adolescents of child bearing potential: being willing and able to use contraceptive methods for the duration of the study and for 30 days after receiving the last dose of the study drug;
* Diffuse body pain that has been present for at least 3 months, and who also have symptoms of fatigue, sleep disturbance, cognitive changes and mood disorder;
* Accompanied by at least one somatic symptoms to variable degree including irritable bowel syndrome, headaches, menstrual pain, lower urinary tract symptoms, myofascial pain, and temporomandibular pain;
* Symptoms cannot be explained by some other illness;
* Physical examination which should be within normal limits except for tenderness on pressure of soft tissues (i.e. tactile hyperalgesia which is increased pain following a painful stimulus)
* Overall body pain average score ≥ 4
* Moderate to severe physical impairment Functional Disability Inventory > 12 points.
* Stable doses of his/her current medication for at least four weeks
* Not having significant changes in their health conditions (PIGS less than 6 points) after 8 weeks of treatment

Exclusion Criteria:

* Be part of other trials;
* Have a specific diagnosis that can explain the symptoms; including rheumatoid arthritis, systemic lupus erythematosus, scleroderma and/or other connective tissue diseases
* Refuse to donate blood sample;
* Not be able to fill electronic records;
* Cognitive impairment interfering with the clinical evaluations;
* Known intolerance or allergies to KF;
* Been under treatment with other mast cell stabilizer agent;
* Seizures history or actual treatment;
* Coagulopathies or chronic thrombocytopenia;
* Atopic dermatitis (eczema) or chronic urticaria (hives)
* Schizophrenia or bipolar disorder
* Elective surgery within the study timeline
* Abnormal labs results (i.e., elevated SGPT and low platelet count, low Hb or Ht) in the last 6 months or in the base line evaluation
* Patients who are pregnant or are breast-feeding;
* Patients who are on oral antidiabetic agents;

Ages: 14 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 44 (Actual)
Dates: Start 2016-12 (Actual); Primary Completion 2020-01 (Actual); Study Completion 2020-01 (Actual)

PRIMARY OUTCOMES:
Patients' Global Impression of Change (PGIC) scale | Baseline versus week 16
  "Since beginning treatment, how would you describe the change (if any) in ACTIVITY LIMITATIONS, SYMPTOMS, EMOTIONS and OVERALL QUALITY OF LIFE related to your painful condition?" (CHOOSE ONE).
  * No change (or condition has got worse)
  * Almost the same, hardly any change at all
  * A little better, but not noticeable change at all
  * Somewhat better, but the change has not made any real difference
  * Moderately better, and a slight but noticeable change
  * Better, and a definite improvement that has made a real and worthwhile difference
  * A great deal better, and a considerable improvement that has made all the difference
  Patients scoring either 6 or 7 on the PGIC scale are categorized as "improved". Patients scoring either 6 or 7 on the PGIC scale are categorized as "improved". We will use this definition as a dichotomous variable.

SECONDARY OUTCOMES:
Pain sensitivity | Baseline versus week 16
  we will use a 0 to 10 numerical ranking scale adapted to RedCap to collect pain intensity ratings. In this scale, '0' means 'no pain at all' and '10' means 'the worst intense pain imaginable'. At baseline, weeks 4, 8, 12 and 16 clinical visits, patients will be asked by the research team to rate their lowest, average, and highest pain intensity for the previous day.
  Intensity of the lowest, average, and highest pain at 'week 16' will be on of the secondary end points of the study.
Proportion of patients with pain sensitivity reduced by half | Baseline versus week 16
  We are also interested in the proportion of patients that show a 50% reduction in their pain intensity after 16 weeks of treatment with KF. Thus, we will assess this proportion also for the lowest, average, and highest pain intensity.
Daily profile of pain index | Across baseline and weeks 4, 8, 12 and 16 will be evaluated
  As patients rate their lowest, average, and highest pain intensity daily on RedCap, they will be prompted to indicate also for how many hours each of these pains lasted. The product of pain intensity by pain duration (in hours) will generate the pain index (Example: pain intensity of 9 with a duration of 6 hours = pain index 54)
Pressure pain sensitivity | Across baseline and weeks 4, 8, 12 and 16 will be evaluated
  Pressure pain thresholds (PPT) will be determined using a digital pressure algometer with a flat round transducer, applied bilaterally at the trapezius muscle and lateral epicondyle. Pressure will be increased at a steady rate of approximately 1 kg/s until the subject indicates that the pressure sensation is perceived as painful sensation (threshold), and the pressure in kg recorded. The first trial at each test site will be considered a practice trial, and will be excluded from data analysis. In subsequent trials, the pressure level at the time the subject indicates to first perceive the pressure sensation to become a painful sensation will be recorded as the threshold estimate. If no response is given at the point the algometer reaches maximum pressure, the maximum value will be used as the threshold value. This procedure will be repeated three times at each test site, and the mean value will be recorded as the subjects threshold.
Functional Disability Inventory | Compare values at baseline, with those of weeks 4, 8, 12 and 16.
  The scale can be completed in person, by mail, or by phone. Scoring: item scores range from 0-4. The total FDI score is a sum of all of the items and can be easily hand scored. Scores range from 0-60, with higher scores indicating greater functional disability. (no/minimal disability 0 -12, moderate disability 13-29, and severe disability >30)
Revised Child Anxiety and Depression Scale (RCADS) | Compare values at baseline, with those of weeks 4, 8, 12 and 16.
  ): is a 47-item scale intended to assess children's report of symptoms corresponding to selected DSM-IV anxiety disorders and depression. The RCADS is a 47-item scale with subscales including: separation anxiety disorder (SAD), social phobia (SP), generalized anxiety disorder (GAD), panic disorder (PD), obsessive compulsive disorder (OCD), and major depressive disorder (MDD). It also yields a Total Anxiety Scale (sum of the 5 anxiety subscales) and a Total Internalizing Scale (sum of all 6 subscales). Recall period for item: one week. Scoring programs are available at www.childfirst.ucla.edu/resources for scoring the RCADS.
Sleep | Compare values at baseline, with those of weeks 4, 8, 12 and 16.
  Pittsburgh Sleep Quality Index (PSQI): 19 items scale assessing sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, use of sleeping medications, and daytime dysfunction. Recall period for item: one month Scoring: Point values of each item in of the seven subscales are summed and then combined as indicated to generate a subscale score. These totals are summed to create the global PSQI score.
Role Functioning | Compare values at baseline, with those of weeks 4, 8, 12 and 16.
  Patients will be asked at each evaluation to quantify the number of days lost because of pain and/or associated symptoms in the previous four weeks. Days of school missed because of medical appointments will not be quantified for the role functioning analysis.
Analgesic medication reduction | Compare baseline with weeks 4, 8, 12 and 16.
  Patients will be allowed to reduce the doses or, eventually, to stop the use analgesic medication under medical supervision if there is a significant reduction in pain intensity (50% reduction in pain intensity rating) or in the associated symptoms
Adverse events | Compare weeks 4, 8, 12 and 16.
  We will use an electronic list of adverse reactions to check for treatment-emergent adverse events. This list was created by us to run on RedCap, based on the list of adverse reactions reported by patients participating in a double-blind, placebo controlled Canadian Multicentre Trial (196 asthmatic children aged 5- 17 years) (Rackham, A. et al. A Canadian multicenter study with Zaditen (ketotifen) in the treatment of bronchial asthma in children aged 5 to 17 years. The Journal of allergy and clinical immunology 84, 286-296 (1989).
RNA expression | Baseline versus week 16
  RNA expression patterns will be compared before and after treatment,

CONTACTS AND LOCATIONS:
Locations (1):
- McGill University Health Centre (MUHC) - Montreal Children's Hospital, Montreal, Quebec, Canada